CLINICAL TRIAL: NCT07148388
Title: Effects and Mechanism of Accelerated Intermittent Theta Burst Stimulation on Neuropathic Pain
Brief Title: Accelerated Intermittent Theta Burst Stimulation (AiTBS)on Neuropathic Pain
Acronym: AiTBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Yan, prof., Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-0669
Record Dates: First submitted 2025-08-04; First posted 2025-08-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-07

CONDITIONS: Neuropathic Pain, Nociceptive Pain
Keywords: AiTBS, rTMS, Neuropathic pain
MeSH Terms: conditions — Neuralgia; Nociceptive Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AiTBS group (Experimental): Eligible patients were receive 5 days of AiTBS on left M1 within 10 days. Clinical and neurophysiological assessments were performed at baseline and after the last sessions.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- 10Hz rTMS (Active Comparator): Patients were assigned to receive 10 consecutive days of classic 10Hz rTMS intervention on left M1. Clinical and neurophysiological assessments were performed at baseline and after the last sessions.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Patients in the AiTBS group received 5 consecutive days of AiTBS treatment, with 6 sessions of iTBS interventions per day (1800 pulses per trial, with a 50-minute interval between trials). Patients in the 10Hz rTMS group received 10 consecutive days of 10Hz rTMS treatment within 10 days, with 1500 pulses per day, totaling 15 minutes.

SUMMARY:
The present study was designed to be the first to evaluate the efficacy of the AiTBS protocol to relieve neuropathic pain in a therapeutic setting, i.e. with repeated stimulation sessions. The investigator directly compared the analgesic efficacy of AiTBS versus conventional 10-Hz rTMS delivered to the left M1. In addition to pain experiences, The investigator examined the effects of intervention on corticospinal excitability that assessed by TMS-EEG. The working hypothesis was that AiTBS would result in larger analgesic and significant cortical excitability changes compared to 10-Hz rTMS.

Eligible patients were randomly assigned to receive either 5 days of AiTBS within 10 days (6 sessions per day) or 10 consecutive days of classic 10Hz rTMS intervention. Clinical and neurophysiological assessments were performed at baseline and after the last sessions.

ELIGIBILITY:
Inclusion Criteria:

* IASP diagnosis of peripheral neuropathic pain;
* At least three months after the onset of pain;
* At least moderate pain intensity (≥ 3 assessed by VAS or NRS);
* 18 years or older;
* Stable medical treatment from 2 weeks before allocation to the end of the trial;
* Willing to receive TMS treatment and capable of fulfilling clinical assessments.

Exclusion Criteria:

* Contradictions to TMS treatment, such as metal implants or seizure;
* Serious psychiatric disorder (Hamilton Depression Rating Scale score ≥ 35 or Hamilton Anxiety Rating Scale score ≥ 29);
* Aphasia or cognitive disorders (Mini mental state examination ≤ 24);
* Severe clinical disorders caused by tumor or other conditions;
* Severe cardiopulmonary dysfunction or extreme weakness;
* History of substance abuse (alcohol, drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group, 1 month after intervention
  It typically consists of a 10-centimeter straight line, with two endpoints representing extreme states of the measured experience. For example, when assessing pain, one end is labeled "0 (no pain at all)" and the other end "10 (worst pain imaginable, unbearable)".
  The individual being evaluated marks a point on the line that corresponds to their current experience. The score is determined by measuring the distance from this mark to the "0" end, converted into a numerical value ranging from 0 to 10 (where each centimeter equals 1 point). Higher scores indicate a stronger intensity of the experience.

SECONDARY OUTCOMES:
short-form McGill Pain Questionnaire (SF-MPQ) | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group, 1 month after intervention
  The Short-Form McGill Pain Questionnaire (SF-MPQ) is a concise, widely used tool designed to assess the nature and intensity of pain in a efficient manner.
  Key Components:
  * Sensory pain descriptors (11 items): These words capture the physical qualities of pain, such as "throbbing," "burning," "aching," and "sharp." Respondents rate each on a scale of 0 (none) to 3 (severe).
  * Affective pain descriptors (4 items): These reflect the emotional aspects of pain, including "tiring," "fearful," "punishing/cruel," and "worrying." They are also rated 0-3.
  * Visual Analog Scale (VAS): A 10-centimeter line with endpoints labeled "no pain" and "worst imaginable pain." Patients mark a point along the line to indicate their pain intensity.
  * Present Pain Intensity (PPI): A 6-point scale (0-5) ranging from "no pain" (0) to "excruciating" (5), used to rate the current level of pain.
7-item pain interference scale of the Brief Pain Inventory (BPI) | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group, 1 month after intervention
  * Items assessed: The 7 items evaluate how pain interferes with:
    * General activity
    * Mood
    * Walking ability
    * Normal work (including both work outside the home and housework)
    * Relationships with others
    * Sleep
    * Enjoyment of life
  * Rating scale: Each item is rated on an 11-point numerical scale (0 = "does not interfere" to 10 = "interferes completely"), based on the past 24 hours.
The Patient Global Impression of Change (PGIC) | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group, 1 month after intervention
  * Single-item structure: It consists of a single question that asks patients to rate how much their condition has changed since a specified baseline (e.g., "Since starting treatment, how would you rate your overall change in pain?").
  * 7-point response scale: Responses range from "very much improved" (score 1) to "very much worse" (score 7), with intermediate options including "much improved," "minimally improved," "no change," "minimally worse," and "much worse."
  * Subjective and holistic: It captures the patient's personal, global judgment rather than focusing on specific symptoms, reflecting their integrated experience of change.
The 17-item Hamilton Depression Rating Scale (HAMD-17) | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group, 1 month after intervention
  It includes 17 items covering core depressive symptoms and related manifestations, mainly involving the following dimensions:
  * Emotional symptoms: Such as depressed mood, feelings of guilt, suicidal ideation, etc.
  * Somatic symptoms: Including difficulty falling asleep, difficulty maintaining sleep, early awakening, reduced work and interests, retardation (psychomotor), agitation (psychomotor), somatic anxiety, gastrointestinal symptoms, general symptoms, sexual symptoms, etc.
  * Other related symptoms: Such as weight loss, insight, delusional or obsessive symptoms, depersonalization or derealization, paranoid symptoms, compulsive symptoms, etc. (Some items vary slightly according to versions, with the core being emotional and somatic manifestations related to depression).
The Beck Depression Inventory-II (BDI-II) | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group, 1 month after intervention
  The Beck Depression Inventory-II (BDI-II) is a widely used self-report questionnaire designed to assess the severity of depressive symptoms in adults and adolescents.
  It consists of 21 items, each describing a specific depressive symptom (e.g., sadness, loss of interest, guilt, fatigue, sleep disturbances, appetite changes).
TMS-EEG | Day1(Baseline), day 5 in AiTBS group, day 10 in 10Hz group
  TMS-EEG (Transcranial Magnetic Stimulation-Electroencephalography) is a combined neuroimaging technique that synchronously uses TMS to non-invasively stimulate specific brain regions and EEG to record the brain's electrical activity responses to this stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No